CLINICAL TRIAL: NCT03782870
Title: Clinical and Echocardiographic Evaluation of Patients With Granulomatosis With Polyangiitis
Brief Title: Cardiovascular Involvement in Patients With Granulomatosis With Polyangiitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: AKBE/130/2018
Record Dates: First submitted 2018-12-13; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Granulomatosis With Polyangiitis; Atherosclerosis; Thrombosis
Keywords: granulomatosis with polyangitis, cardiac involvement
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Atherosclerosis; Thrombosis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echocardiography, lab tests

SUMMARY:
Granulomatosis with polyangiitis (GPA) is one of antineutrophil cytoplasmic autoantibody (ANCA) - associated vasculitis. Inflammation-induced thrombosis is considered to be a feature of systemic autoimmune diseases. GPA usually involves the upper and lower respiratory tract and renal systems, where necrotizing glomerulonephritis and pulmonary capillaritis are often detected. However, it may also affect other organ systems. Cardiac involvement in GPA occurs in approximately 6% to 44% of cases and is secondary to necrotizing vasculitis with granulomatous infiltrates. Cardiac involvement is an independent predictor of mortality in GPA patients. In this prospective cohort study, consecutive GPA patients who were hospitalized in the Department of Family Medicine, Internal and Metabolic Diseases at the Medical University of Warsaw in Poland are included. In all patients echocardiography and laboratory tests are perform.

DETAILED DESCRIPTION:
Granulomatosis with polyangiitis (Wegener's; GPA) is an antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV), which also includes microscopic polyangiitis and eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome). GPA is characterized by granulomatous inflammation and necrotizing vasculitis predominantly affecting small- to medium-sized blood vessels and the presence of ANCA directed to specific antigens, particularly proteinase 3 (PR3-ANCA) and myeloperoxidase (MPO-ANCA). The destructive inflammatory processes of GPA have a predilection for the upper and lower airways and the kidneys, but any organs can be affected. An increased incidence of various cardiovascular events has been demonstrated among GPA patients. Cardiac involvement is also an independent predictor of mortality in GPA patients. In this prospective cohort study, consecutive GPA patients who are hospitalized in the Department of Family Medicine, Internal and Metabolic Diseases at the Medical University of Warsaw in Poland are included. All patients are diagnosed with GPA according to current guidelines. Patients are entered into the study at the time point when a new diagnosis of GPA was established and received initial treatment at our centre. Data collection included a full interim medical history, physical examination, laboratory studies and review of adverse events. Additionally, in all patients an echocardiography is performed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Granulomatosis with polyangitis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed Granulomatosis with polyangitis who received initial treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-02-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
death from any cause | from date of randomization until the death from any cause, up to december 2018
  death

SECONDARY OUTCOMES:
coronary artery disease | from date of randomization until the date of first documented coronary artery disease episodes up to december 2018
  coronarography
stroke | from date of randomization until the date of documented stroke, up to december 2018
  CT scan
deep vein thrombosis | from date of randomization until the date of documented deep vein thrombosis, up to december 2018
  Ultrasonography of the lower extremity veins

CONTACTS AND LOCATIONS:
Overall Officials: Anna Borowiec, PhD, Study Chair — Warsaw University of Medicine
Locations (1):
- Department of Family Medicine, Internal and Metabolic Diseases, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided